CLINICAL TRIAL: NCT04588051
Title: A Phase II Clinical Trial to Study the Efficacy of Cabozantinib in Patients with Hepatocellular Carcinoma Refractory to Checkpoint Inhibitors
Brief Title: Cabozantinib in Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Chan Lam (Other)
Responsible Party: Sponsor-Investigator, Stephen Chan Lam, Associate Professor, Department of Clinical Oncology, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC063
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: HCC
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib (Experimental)
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — 60mg daily

SUMMARY:
There have been lack of clinical studies on the role of drug treatment in patients who develop progressive disease with immune checkpoint inhibitors. Amongst HCC patients who become intolerant or refractory to sorafenib, cabozantinib has been shown by phase III clinical trial (CELESTIAL) to prolong the overall survival of patients, as compared to placebo. It is expected more patients will be treated with immune checkpoint inhibitors in future, hence it is clinically important to study the efficacy and toxicity of cabozantinib after treatment with immune checkpoint inhibitors.

Further, both MET activation and upregulation of regulatory T cells are implicated in resistance mechanism to immune checkpoint inhibitors. Immuno-modulatory effects of cabozantinib have been described in vitro and in murine models for several cancers. Moreover, cabozantinib appears to exert its effect on regulatory T cells (Tregs) via the HGF/c-Met pathway, where this receptor signaling cascade mediates multiple immune cell functions. HGF was shown to suppress DC function and in turn induce Tregs (CD4+ CD25+ FoxP3) in a murine central nervous system (CNS) autoimmunity model. HGF cultured monocytes differentiate into monocytic cells that produce soluble factors that favor immune suppressive conditions ideal for tumor progression. Above immunomodulatory effects could enable cabozantinib to reverse the immunosuppressive phenotype in patients after failure with immune checkpoint inhibitors.

The starting dose of cabozantinib of 60mg once daily in the current study is chosen in accordance with approved dose by FDA for treatment of advanced HCC

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC according to AASLD guidelines
2. Disease that is not amenable to a curative treatment (e.g. surgery, transplant, radiofrequency ablation)
3. Prior treatment with immune check-point inhibitor (including anti-PD1, anti-CTLA4, anti-PD1 plus anti-CTLA4, or above agents plus other targeted agents)
4. For patients who stop immune check-point inhibitor due to progressive disease, the duration of immune check-point inhibitor must be 8 weeks or longer
5. Recovery to ≤ Grade 1 from toxicities related to any prior treatments, unless the adverse events are clinically nonsignificant and/or stable on supportive therapy
6. Life expectancy of 12 weeks or longer
7. Age ≥ 18 years old
8. ECOG performance status of 0, 1 or 2
9. Adequate hematological function

   1. Absolute neutrophil count (ANC) ≥ 1.2 x109/L
   2. Platelets ≥ 60 x 109/L
   3. Hemoglobin ≥ 8g/dL
10. Adequate renal function

    1. serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockroft-Gault equation) AND
    2. urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1 g
11. Child-Pugh Score of A5 or 6
12. Total bilirubin ≤ 2 mg/dL (≤ 34.2 μmol/L)
13. Serum albumin > 2 g/dL (> 20 g/L)
14. Alanine aminotransferase (ALT) < 3.0 upper limit of normal (ULN)
15. Hemoglobin A1c (HbA1c) ≤ 8%
16. Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
17. Capable of understanding and complying with the protocol requirements and signed informed consent
18. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment
19. Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Prior cabozantinib treatment
3. More than two lines of systemic therapy (i.e. cabozantinib must be either 2nd line or 3rd line systemic treatment)
4. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before randomization.
5. Concurrent steroid use of prednisolone >10mg once daily
6. Presence of thrombosis or tumor invasion in inferior vena cava
7. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low dose LMWH are permitted.
8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders including i. Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias ii. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment iii. Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months iv. Thromboembolic event within 3 months. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumour are eligible b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation/bleeding: i. Tumours invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months
9. Major surgery within 2 months before randomization. Complete healing from major surgery must have occurred 1 month before randomization. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before registration. Subjects with clinically relevant co d. Cavitating pulmonary lesion(s) or endobronchial disease
10. Lesion invading a major blood vessel (eg, pulmonary artery or aorta)
11. Clinically significant bleeding risk including the following within 3 months of registration: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
12. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding are excluded with the following clarification: subjects with history of prior variceal bleeding must have been treated with adequate endoscopic therapy without any evidence of recurrent bleeding for at least 6 months prior to study entry and must be stable on optimal medical management (e.g. non-selective beta blocker, proton pump inhibitor) at study entry.
13. Moderate or severe ascites (Radiologically detected but clinically insignificant ascites is allowed)
14. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 21 days of registration Note: If the QTcF is > 500 ms in first ECG, a total of 3 ECGs should be performed. If the average of these 3 consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
15. Previously identified allergy or hypersensitivity to components of the study treatment formulations
16. Pregnant or lactating females
17. Diagnosis of another malignancy within 2 years before randomization, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
18. Other clinically significant disorders that are judged by investigators to be unsuitable for the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression-free survival (PFS) | 1 year

SECONDARY OUTCOMES:
Median Overall survival (OS) | 1 year
Survival rate at 1-year | 1 year
Median time-to-progression | 1 year
Radiological response rate (RR) according to RECIST 1.1 | 1 year
Radiological disease control rate (DCR) according to RECISIT 1.1 | 1 year
Rate of adverse events according to CTCAE v5.0 | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong
- ASAN Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SL, Ryoo BY, Mo F, Chan LL, Cheon J, Li L, Wong KH, Yim N, Kim H, Yoo C. Multicentre phase II trial of cabozantinib in patients with hepatocellular carcinoma after immune checkpoint inhibitor treatment. J Hepatol. 2024 Aug;81(2):258-264. doi: 10.1016/j.jhep.2024.03.033. Epub 2024 Apr 1. PMID 38570034